CLINICAL TRIAL: NCT04877496
Title: Registry Study for COVID19 Vaccination Efficacy in Patients With a Treatment History of Rituximab.
Brief Title: Responses to COVID19 Vaccination in Patients With a Treatment History of Rituximab.
Acronym: RituxiVac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 4749
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: COVID19 Vaccination; Rituximab; Immunosuppression
Keywords: B-cells; T-cells; COVID19 vaccine; SARS-CoV2; Rituximab
MeSH Terms: interventions — F-Box-WD Repeat-Containing Protein 7

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunocompetent controls: Participants aged at least 18 years, no history of COVID19, no history of anti-CD20 treatment
  Interventions: Biological: Completion of COVID19 vaccine at least 4 weeks ago
- Patients with a treatment history of rituximab: Participants aged at least 18 years, no history of COVID19, history of at least 1 dose of anti-CD20 treatment received since 01/01/2010
  Interventions: Drug: History of exposure to anti-CD20 treatment since 01/01/2010; Biological: Completion of COVID19 vaccine at least 4 weeks ago

INTERVENTIONS:
Drug: History of exposure to anti-CD20 treatment since 01/01/2010 — Intravenous treatment history of anti-CD20 treatment since 01/01/2010
  Groups: Patients with a treatment history of rituximab
Biological: Completion of COVID19 vaccine at least 4 weeks ago — Completion of COVID19 vaccination course at least 4 weeks ago.

SUMMARY:
Patients with treatment history of rituximab since 01.01.2019 and immunocompetent volunteers will be contacted to give a blood sample after their COVID19 vaccination, and in a subset also before vaccination. Immune responses of antibodies and SARS-CoV2-specific T-cells to the vaccination will be quantified and the rituximab effect on COVID19 vaccine-induced immune responses is analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were treated with anti-CD20 treatment since 01.01.2010
2. Patients who received a COVID19 vaccination (completion of all required doses) until target date (initial target: 30.05.21, but can be delayed to 30.06.21, 30.07.21 or 30.08.21 in case of insufficient enrollment)
3. Volunteers without a history of anti-CD20 treatment exposure
4. All: written informed consent.

Exclusion Criteria:

Exclusion criteria for patients (any of the following)

1. Patients aged 18 years and younger at time of study enrollment and/or
2. Pregnant or lactating women at time of study enrollment and/or
3. Patients who do not provide written informed consent and/or
4. Patients who have previously had a COVID19 infection (self-reported COVID19 disease, positive PCR or serology)
5. Patients who are in a dependency relationship with the study personnel (hierarchical, social)

Exclusion criteria for volunteers (any of the following)

1. Volunteers aged 18 years and younger at time of study enrollment and/or
2. Pregnant or lactating women at time of study enrollment and/or
3. Volunteers who do not provide informed consent and/or
4. Volunteers who suffer from an active autoimmune disease, active cancer, immunosuppressive therapy, history of anti-CD20 treatment and/or
5. Volunteers who have previously had a COVID19 infection (self-reported COVID19 disease, positive PCR or serology)
6. Volunteers who did not complete their COVID19 vaccination
7. Volunteers who are in a dependency relationship with the study personnel (hierarchical, social)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-represented gender.
Study Population: Participating Centers / Participating Departments: all at Bern University Hospital Insel)
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response to SARS-CoV2 spike protein | At least 4 weeks after completion of COVID19 vaccination
  Percentage of all patients developing IgG antibodies against SARS-CoV2 spike protein that is comparable to the immunological response in immunocompetent controls (-2 standard deviations of mean)

SECONDARY OUTCOMES:
Correlation of IgG antibodies against SARS-CoV2 with age, history, co-medication and biomarkers of immunocompetence | At least 4 weeks after completion of COVID19 vaccination
  Multivariable regression models for IgG antibodies against SARS-CoV2 with age, history, co-medication and biomarkers of immunocompetence as confounding variables.
Correlation of IgG antibodies against SARS-CoV2 with time interval since last dose of rituximab | At least 4 weeks after completion of COVID19 vaccination
Correlation of IgG antibodies against SARS-CoV2 with cumulative dose of rituximab received. | At least 4 weeks after completion of COVID19 vaccination
T cell anti-SARS-CoV2 response after COVID19 vaccination | At least 4 weeks after completion of COVID19 vaccination
Correlation between IgG antibodies against SARS-CoV2 and B-cell counts, T-cell counts and total immunoglobulin levels | At least 4 weeks after completion of COVID19 vaccination
  Multivariable regression models for IgG antibodies against SARS-CoV2 with B-cell counts, T-cell counts and total immunoglobulin levels as confounders.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sidler, MD PhD, Principal Investigator — University Hospital Bern, Department of Nephrology and Hypertension
Locations (1):
- University Hospital Bern Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sidler D, Born A, Schietzel S, Horn MP, Aeberli D, Amsler J, Moller B, Njue LM, Medri C, Angelillo-Scherrer A, Borradori L, Seyed Jafari SM, Radonjic-Hoesli S, Chan A, Hoepner R, Bacher U, Mani LY, Iype JM, Suter-Riniker F, Staehelin C, Nagler M, Hirzel C, Maurer B, Moor MB. Trajectories of humoral and cellular immunity and responses to a third dose of mRNA vaccines against SARS-CoV-2 in patients with a history of anti-CD20 therapy. RMD Open. 2022 Mar;8(1):e002166. doi: 10.1136/rmdopen-2021-002166. PMID 35361691
- [Derived] Moor MB, Suter-Riniker F, Horn MP, Aeberli D, Amsler J, Moller B, Njue LM, Medri C, Angelillo-Scherrer A, Borradori L, Radonjic-Hoesli S, Seyed Jafari SM, Chan A, Hoepner R, Bacher VU, Mani LY, Iype JM, Hirzel C, Maurer B, Sidler D. Humoral and cellular responses to mRNA vaccines against SARS-CoV-2 in patients with a history of CD20 B-cell-depleting therapy (RituxiVac): an investigator-initiated, single-centre, open-label study. Lancet Rheumatol. 2021 Nov;3(11):e789-e797. doi: 10.1016/S2665-9913(21)00251-4. Epub 2021 Sep 7. PMID 34514436